CLINICAL TRIAL: NCT03290053
Title: Contrast Enhanced Sonothrombolysis and Sonolysis in Stroke - a Swedish Study (CE-5S)
Acronym: CE-5S
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor inclusion rate & lack of funding
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE-5S
Record Dates: First submitted 2017-09-14; First posted 2017-09-21 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2017-11

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — contrast agent BR1; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CE-5S A: Treatment arm (Experimental): Gets thrombolysis, transcranial ultrasound on the flow limitation and SonoVue infusion
  Interventions: Drug: SonoVue; Procedure: Transcranial Ultrasound
- CE-5S A: Control arm (Sham Comparator): Gets thrombolysis, sham transcranial ultrasound and placebo (NaCl) infusion
  Interventions: Drug: Sodium chloride; Procedure: Sham Transcranial Ultrasound
- CE-5S B: Treatment arm (Experimental): Gets NO thrombolysis (due to contraindications), transcranial ultrasound on the flow limitation and SonoVue infusion
  Interventions: Drug: SonoVue; Procedure: Transcranial Ultrasound
- CE-5S B: Control arm (Sham Comparator): Gets NO thrombolysis (due to contraindications), sham transcranial ultrasound and placebo (NaCl) infusion
  Interventions: Drug: Sodium chloride; Procedure: Sham Transcranial Ultrasound

INTERVENTIONS:
Drug: SonoVue — SonoVue-infusion over 1 hour
  Arms: CE-5S A: Treatment arm; CE-5S B: Treatment arm
Drug: Sodium chloride — Placebo
  Arms: CE-5S A: Control arm; CE-5S B: Control arm
Procedure: Transcranial Ultrasound — Transcranial ultrasound aimed at the blockage
  Arms: CE-5S A: Treatment arm; CE-5S B: Treatment arm
Procedure: Sham Transcranial Ultrasound — Placebo - machine is attached, but not active
  Arms: CE-5S A: Control arm; CE-5S B: Control arm

SUMMARY:
Patients with acute ischemic stroke in anterior circulation within 4,5 hours of symptom onset, has a bone window and Trombolysis In Brain Ischemia (TIBI) <=4 in a relevant artery eligible. Both patients receiving thrombolysis and those who do not due to contraindications such as anticoagulation or recent surgery are enrolled, but into different study arms (CE-5S A for thrombolysis and B for non-thrombolysis); the decision to treat with thrombolysis or not is done according to clinical routine.

All included patients are randomized to receive transcranial ultrasound and SonoVue-infusion or sham-ultrasound and placebo; i.e. in CE-5S A, contrast enhanced sonothrombolysis is compared to thrombolysis and in CE-5S B, contrast enhanced sonolysis is compared with conservative management.

Main outcome is improvement in National Institute of Health Stroke Scale (NIHSS) at 24 hours compared to baseline. Main safety outcome is symptomatic intracerebral haemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years with acute ischaemic stroke in the anterior circulation, who has given written consent for his/her participation to the study.
* Remaining neurological deficit that is ≥1 NIHSS points, sufficient to warrant treatment with tPA (not taking possible contraindications into account) and is severe enough that possible improvement is clearly analysable
* Treatment <4½ hours of symptom onset or of waking up in the morning with symptoms
* Sufficient bone window for acceptable or better acquisition of flow information with ultrasound with TIBI ≤ 4 in the symptomatic artery
* In cases with women of Childbearing Capacity (WOCBC): Only if willing to comply with effective contraception methods during the course of the trial. Acceptable methods are such as oral contraceptives, contraceptive patches, contraceptive implant, vaginal contraceptive, double-barrier methods (for example, condom and spermicide), intrauterine device (IUD), hormonal IUD

Exclusion Criteria:

* Patients with premorbid modified Rankin Scale (mRS) score ≥3;
* Patients for whom a complete NIHSS cannot be obtained;
* Hemiplegic migraine with no arterial occlusion on baseline Computed Tomography of brain (CT);
* Seizure at stroke onset and no visible occlusion on baseline CT;
* Intracranial haemorrhage on baseline CT;
* Clinical presentation suggesting subarachnoid haemorrhage even if baseline CT is normal;
* Large areas of hypodense ischaemic changes on baseline CT;
* Pregnancy or breast-feeding, pericarditis; sepsis; any other serious medical illness likely to interact with treatment; confounding pre-existent neurological or psychiatric disease; unlikely to complete follow-up; any investigational drug <14 days;
* Inability to provide informed consent sufficiently clearly that the study physician can be convinced that informed consent has been given by the patient - such as severe aphasia or coma.

Specific sonothrombolysis exclusion criteria

* known hypersensitivity/allergy to SonoVue;
* recent or unstable coronary ischemia or resting angina <7 days;
* acute cardiac insufficiency, cardiac insufficiency class III/IV; serious cardiac arrhythmias;
* any right-left-shunt; severe pulmonary hypertension; uncontrolled hypertension;
* moderate to severe Chronic Obstructive Pulmonary Disease (COPD; baseline O2 saturation <80%);
* acute respiratory distress syndrome (ARDS);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Early clinical Outcome defined as change in NIHSS at 24 hours. | 24 hours
  Change in National NIHSS at 24 hours. Defined reaching of primary endpoint is post-treatment 0 Points and/or improves with >=4 Points compared to pre-treatment.

SECONDARY OUTCOMES:
Safety: Symptomatic Cerebral Hemorrhage (sICH) | 24-36 hours
  Assessed with routine post-treatment CT head and requires an accompanied >=4 Points worsening on NIHSS.
Long term outcome defined as residual handicap at Three months | 90 days
  90-days modified Rankin Scale (mRS) reaching 0-1.

CONTACTS AND LOCATIONS:
Overall Officials: Elias Johansson, MD, PhD, Principal Investigator — Umeå University
Locations (1):
- University Hospital, Umeå, Västerbotten County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided